CLINICAL TRIAL: NCT01382251
Title: Functional Recovery and Caregiver Burden Following Surgery in the Elderly
Acronym: FOCUS
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Anesthesiologists' Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2009390-01H
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Activities of Daily Living; Caregivers; Ambulatory Surgical Procedures
Keywords: Activities of Daily Living; Caregivers; Ambulatory Surgical Procedures

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient: Patients undergoing ambulatory surgery
- Caregiver: Spouse, family members, or friends identified as the patient's primary source of support in the community.

SUMMARY:
The purpose of this study is to assess the functional recovery of older ambulatory surgical patients and the impact of the current model of care on the caregivers of these patients. This study will provide unique insight into the challenges patients and their families face following surgery.

The primary objective of this study is to:

1. Assess the impact of ambulatory surgery on functional capacity as assessed by the Système de Mesure de l'Autonomie Fonctionnelle (SMAF) one week and one month following surgery in a population of surgical patients 65 years of age and older.

   Secondary objectives are to determine if:
2. Changes in the patient's functional capacity result in increased burden of care as assessed by the Zarit Burden Interview (ZBI) in the patient's primary caregiver.
3. Changes in functional capacity are correlated with decrements in quality of life as assessed by the Short Form 12 (SF12).
4. Changes in functional capacity are correlated with inadequate postoperative analgesia as assessed by the Brief Pain Inventory (BPI).

ELIGIBILITY:
Inclusion Criteria:

Patients

* aged 65 years and older
* elective surgery with a planned discharge to the community on the day of the surgical procedure.
* Eligible surgical procedures include: inguinal herniorrhaphy, ventral herniorrhaphy, laparoscopic cholecystectomy,laparoscopic salpingoophorectomy, urethropexy, cystocoele/rectocoele repair, vaginal hysterectomy, arthroscopic debridement (knee, hip, shoulder), arthroscopic repair (knee, hip, shoulder), removal of hardware from lower extremity, foot surgery, and lumbar discectomy.

Caregiver

- spouses, family members, or friends identified as the patient's primary source of support in the community.

Exclusion Criteria:

Patients

* Reside in a nursing home providing professional support services;
* Are unable to complete the study instruments due to cognitive (MMSE <24) or physical impairment;
* Are unable to speak English or French

Caregiver

* Professional caregivers (nurse, personal care assistant, etc) hired to care for the patient;
* Unable to complete the study instruments due to physical impairment;
* Unable to Speak English or French

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing ambulatory surgery and their primary caregivers
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Bryson, FRCPC, Principal Investigator — Department of Anesthesiology, The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Bryson GL, Clavel NA, Moga R, Power B, Taljaard M, Nathan HJ. Patient function and caregiver burden after ambulatory surgery: a cohort study of patients older than 65. Can J Anaesth. 2013 Sep;60(9):864-73. doi: 10.1007/s12630-013-9982-y. Epub 2013 Jun 15. PMID 23771742
- [Derived] Bryson GL, Mercer C, Varpio L. Patient and caregiver experience following ambulatory surgery: qualitative analysis in a cohort of patients 65 yr and older. Can J Anaesth. 2014 Nov;61(11):986-94. doi: 10.1007/s12630-014-0229-3. Epub 2014 Sep 9. PMID 25200593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients > 65 yrs scheduled to undergo elective ambulatory orthopedic or peritoneal surgeries were assessed for eligibility. Each patient must have a partner or adult descendant as primary caregiver. Patient-caregiver dyads were approached in the pre-admission unit. Screening began on 2010-07-01 and the final assessment was completed on 2012-01-04.
Period: Overall Study
Arm/Group | Ambulatory Surgery Patients | Ambulatory Surgery Caregivers
Started | 123 | 123
Completed | 102 | 102
Not Completed | 21 | 21
Not completed — Surgeries cancelled or delayed | 16 | 16
Not completed — Lost to Follow-up | 4 | 4
Not completed — Contacted after study closed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Demographic characteristics shown for those patients and caregivers completing study
Groups:
- Ambulatory Surgery Patients: Only patients with caregivers were recruited
- Ambulatory Surgery Caregivers: Caregivers were recruited with the patients receiving surgery
- Total: Total of all reporting groups
Arm/Group | Ambulatory Surgery Patients | Ambulatory Surgery Caregivers | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 30 | 30
  >=65 years | 102 | 72 | 174
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 48 | 47 | 95
Region of Enrollment [Number; unit: participants]
  Canada | 102 | 102 | 204

OUTCOME MEASURES:

1. Primary Outcome: Functional Autonomy Measurement System (SMAF)
Description: 29-item scale, each item graded on a four-point scale. 0= independent, 1= needs supervision,2 = needs help, 3 = dependent. Total score ranges from 0 to 87 with higher scores indicating increased disability
Time Frame: Baseline, one week, and one month following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambulatory Surgery Patients | Ambulatory Surgery Caregivers
Number analyzed (Participants) | 102 | 102
units on a scale
  Baseline | 4.0 (5.9) | 2.0 (2.9)
  One Week Post-op | 10.9 (7.6) | NA (NA) — Did not undergo surgery therefore no anticipated change in function
  One Month Post-op | 6.7 (7.2) | NA (NA) — Did not undergo surgery therefore no anticipated change in function

2. Secondary Outcome: Zarit Burden Interview (ZBI)
Description: A 22-item questionnaire in which subjects rate how often they experience negative feelings associated with caregiving. Each item rated on a 5 point scale anchored at 0 for "never" and 4 for "nearly always." Scores range from 0-88 with higher scores indicating increased burden of care.
Time Frame: Baseline, one week, and one month following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambulatory Surgery Patients | Ambulatory Surgery Caregivers
Number analyzed (Participants) | 0 | 102
units on a scale
  Baseline |  | 9.3 (9.9)
  One Week Post-op |  | 8.9 (9.8)
  One Month Post-Op |  | 8.6 (10.6)

3. Secondary Outcome: Short Form 12
Description: A validated measure of health related quality of life comprised of 12 questions regarding participant experience over the preceding week. Generate Physical And Mental Component scores ranging from 0-100 with higher scores indicating better quality of life.
Time Frame: Baseline, one week, and one month following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambulatory Surgery Patients | Ambulatory Surgery Caregivers
Number analyzed (Participants) | 102 | 102
units on a scale
  Mental Component Score (Baseline) | 55.3 (7.5) | 55.9 (6.6)
  Mental Component Score (One Week Post-op) | 54.9 (8.8) | 54.4 (9.0)
  Mental Component Score (One Month Post-Op) | 56.2 (7.8) | 54.8 (8.0)
  Physical Component Score (Baseline) | 43.4 (12.7) | 50.5 (7.9)
  Physical Component Score (One Week Post-op) | 35.1 (10.3) | 51.2 (8.4)
  Physical Component Score (One Month Post-op) | 42.7 (11.4) | 51.3 (8.9)

4. Secondary Outcome: Brief Pain Inventory (BPI) Functional Interference Score.
Description: Comprised of seven questions in which the subject is asked to describe the extent to which pain interferes with activity. Scores are anchored at 0 for "does not interfere" and 10 for "completely interferes." The seven resulting scores are averaged and reported as a single value (0 - 10) with higher scores indicating greater interference with function.
Time Frame: Baseline, one week, and one month following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambulatory Surgery Patients | Ambulatory Surgery Caregivers
Number analyzed (Participants) | 102 | 0
units on a scale
  Baseline | 1.8 (2.4) |
  One Week Post-op | 2.1 (2.1) |
  One Month Post-op | 1.2 (1.7) |

ADVERSE EVENTS:
Time Frame: 30 days following surgery
Description: Adverse event data not collected on caregivers as they did not undergo surgery.
Arm/Group | Ambulatory Surgery Patients
Serious Adverse Events (participants affected / at risk) | 4/102
Other Adverse Events (participants affected / at risk) | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambulatory Surgery Patients (N=102)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Uncontrolled Pain (Injury, poisoning and procedural complications) | 1 (1)
Small Bowel Perforation (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Single center, relatively infrequent assessment, assessment of caregiver burden limited to primary caregiver, majority of caregivers were not employed outside the home.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No